CLINICAL TRIAL: NCT00617253
Title: An Open Label, Dose Escalation Safety and Tolerability Trial of the Combination of s.c. Recombinant Human IL-21 (rIL-21) and Sunitinib (Phase 1) Followed by an Open Label Stratified Randomized 2-arm Trial of rIL-21 Plus Sunitinib Versus Sunitinib Alone (Phase 2a) in Subjects With Stage IV Renal Cell Carcinoma
Brief Title: Combination of Recombinant Human IL-21 (rIL-21) and Sunitinib in Stage IV Renal Cell Carcinoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN028-1642; 2006-005751-16 (EudraCT Number)
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Cancer; Renal Cell Carcinoma
MeSH Terms: conditions — Neoplasms; Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental)
  Interventions: Drug: recombinant interleukin-21; Drug: sunitinib
- B (Experimental)
  Interventions: Drug: sunitinib; Drug: recombinant interleukin-21
- C (Experimental)
  Interventions: Drug: sunitinib; Drug: recombinant interleukin-21
- D (Experimental)
  Interventions: Drug: sunitinib; Drug: recombinant interleukin-21

INTERVENTIONS:
Drug: recombinant interleukin-21 — 3 mcg/kg, s.c. injection
  Other Names: NN028, rIL-21
  Arms: A
Drug: sunitinib — Hard gelatine capsules, 12.5 mg
  Other Names: Sutent®
Drug: recombinant interleukin-21 — 10 mcg/kg, s.c. injection
  Other Names: NN028, rIL-21
  Arms: B
Drug: recombinant interleukin-21 — 30 mcg/kg, s.c. injection
  Other Names: NN028, rIL-21
  Arms: C
Drug: recombinant interleukin-21 — 100 mcg/kg, s.c. injection
  Other Names: NN028, rIL-21
  Arms: D

SUMMARY:
This phase 1/2a trial is conducted in Europe. The first part of the trial is a dose escalation safety trial determining the maximum tolerated dose of rIL-21 when administered in combination with sunitinib.

The second part, scheduled to start in September 2008, is a randomised 2-arm trial comparing the anti-tumour effect of rIL-21 plus sunitinib with sunitinib alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified and surgically incurable stage IV Renal Cell Carcinoma
* ECOG performance status of 0 or 1 (i.e. good performance status)
* Life expectancy of at least 3 months

Exclusion Criteria:

* Prior systemic therapy for metastatic disease
* Radiotherapy within the last 4 weeks prior to start of treatment
* Receipt of any investigational drug within 3 months of starting treatment
* History of any other active malignancy within five years prior to enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-07-12 (Actual); Primary Completion 2008-06-30 (Actual); Study Completion 2008-06-30 (Actual)

PRIMARY OUTCOMES:
Toxicity according to CTCAE version 3.0 | For the duration of the trial

SECONDARY OUTCOMES:
Pharmacokinetics | For the duration of the trial
rIL-21 antibodies | For the duration of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (5):
- Germany (3):
  - Novo Nordisk Investigational Site, Frankfurt
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Hanover
- Netherlands (2):
  - Novo Nordisk Investigational Site, Amsterdam
  - Novo Nordisk Investigational Site, Nijmegen

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com